CLINICAL TRIAL: NCT06090981
Title: Early Bolus Surfactant Replacement Therapy Versus Standard Care in Term (>=37 Weeks) Neonates With Actant Replacement Therapy Versus Standard Care in Term Neonates With Meconium Aspiration Syndrome: An Open Label Randomized Control Trial
Brief Title: Early Bolus Surfactant Replacement Therapy Versus Standard Care in Term Neonates With Meconium Aspiration Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Dr. Sushma Nangia, Director Professor & Head, Neonatology, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LHMC/IEC/2021/03/69
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Meconium Aspiration Syndrome; Surfactant Dysfunction
MeSH Terms: conditions — Meconium Aspiration Syndrome; Surfactant Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early bolus surfactant replacement therapy (Experimental): Neonates randomized to this group will receive early bolus surfactant replacement therapy within 2hr of life
  Interventions: Drug: Bovine surfactant
- Standard care (No Intervention): Neonates randomized to this group will be managed as per standard protocol in the neonatal unit.

INTERVENTIONS:
Drug: Bovine surfactant — Dose of surfactant: 4ml/kg Type of surfactant: 4ml/kg
  Arms: Early bolus surfactant replacement therapy

SUMMARY:
The objective of the study is to compare the total duration of respiratory support in term neonates (≥37weeks) with meconium aspiration syndrome, who are provided early(≤2hr) bolus surfactant therapy versus standard care.

DETAILED DESCRIPTION:
Enrolled participants will be randomly assigned to one of two study groups: 1. early(≤2hr) bolus surfactant replacement therapy or 2. standard care

Intervention group: The neonates enrolled in this group will receive early bolus surfactant replacement therapy within 2hr of life.

Control group: The neonates enrolled in this group will receive standard care according to standard unit protocol

ELIGIBILITY:
Inclusion Criteria:

* Gestation age ≥ 37 week
* Cephalic presentation
* Singleton pregnancy
* Age < 2 hours
* Baby delivered through meconium stained amniotic fluid
* Presence of respiratory distress (DOWNE's score ≥4)

Exclusion Criteria:

* Major congenital malformation
* Antenatal diagnosed CHD
* Hydrops fetalis
* Air leaks before enrolment

Ages: 30 Minutes to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Duration of Total respiratory support | Birth to 28 days
  Combined duration of invasive + non invasive ventilation

SECONDARY OUTCOMES:
Severity of respiratory distress | Birth to 28 days
  The severity of respiratory distress will be assessed using Downe's score. These parameters will be documented hourly within first 2 hours before surfactant replacement and in post lavage unto first 24 hrs, 2 hourly unto 48 hrs, and 4 holy thereafter till cessation of respiratory distress
Proportion of neonates requiring mechanical ventilation | Birth to 28 days
  The babies will be assessed for the need for mechanical ventilation as per standard protocol
Proportion of neonates requiring Non Invasive Ventilation | Birth to 28 days
  The babies will be assessed for the need for non invasive ventilation as per standard protocol
Duration of Mechanical Ventilation | Birth to 28 days
  Total duration of Mechanical Ventilation in days
Duration of oxygen therapy | Birth to 28 days
  The duration of oxygen therapy, mode of delivery, Fio2 and flow rates will be documented hourly within first 2 hours before surfactant replacement and in post lavage unto first 24 hrs, 2 hourly unto 48 hrs, and 4 holy thereafter till cessation of respiratory distress
Complications | Birth to 28 days
  Incidence of PPHN, Pneumothorax, HIE, sepsis, airlocks,
Mortality | Birth to 28 days
  All cause mortality
Duration of hospital stay | Birth to 28 days
  Total duration of hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MD, DM (Neo), Study Chair — Lady Hardinge Medical College, New Delhi, India
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India